CLINICAL TRIAL: NCT02844868
Title: Evaluation of the Observance and the Tolerance of a Motor Training Program Combining With Repetitive tDCS Sessions on Walking Performance of Hemiplegic Stroke Patients at the Subacute Stage Post Stroke. ESTIMAH Study
Brief Title: Evaluation of the Observance and the Tolerance of a Motor Training Program
Acronym: ESTIMAH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1608113; 2016-A01249-42 (Other: ANSM)
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Hemiplegia; Stroke
Keywords: stroke; hemiplegia; transcranial direct current stimulation (tDCS); rehabilitation; lower extremity; gait training
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): During the first 20 min of training program, patient will have active tCDS (2 mA )
  Interventions: Device: Active tDCS
- sham tDCS (Sham Comparator): During the first 20 min of training program, patient will have sham tCDS
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — During the first 20 min of training program, patient will have active tCDS : the patient received a 2 mA anodal tDCS over the lower limb ipsilesional motor area. The anodal electrode was positioned on the hotspot previously identified with TMS. The cathode was placed above the contralesional orbit.
  Arms: Active tDCS
Device: Sham tDCS — During the first 20 min of training program, patient will have sham tCDS : the patient received a 2 mA anodal tDCS (only during the first and the last 30 seconds of the stimulation) and then, patient will have sham tDCS. The anodal electrode was positioned on the hotspot previously identified with TMS. The cathode was placed above the contralesional orbit.
  Arms: sham tDCS

SUMMARY:
Transcortical direct current stimulation (tDCS) is an emerging technique in the rehabilitation of hemiplegic patients after stroke.

This study aims to assess the observance and the tolerance of repeated tDCS stimulation over the primary motor cortex of the lower limb coupled to a motor training program, among hemiplegic patients at the sub-acute stage. This is a prospective, randomized, double-blind, study with two parallel groups of 15 subjects each. The study will analyze first, the patient's observance considered good if 75% of the patients completed the entire protocol duration and the tolerance through a questionnaire. The secondary end point will try to estimate, if possible, the effect size of the walking performance measured with the six-minute walk test and aerobic performance measured with VO2peak of this training program compared to the same program combine with placebo stimulations. These evaluations are performed before, during and after the rehabilitation program.

DETAILED DESCRIPTION:
During the initial 20 min of each session, the patient received a 2 mA anodal tDCS over the lower limb ipsilesional motor area. The anodal electrode was positioned on the hotspot previously identified with TMS. The cathode was placed above the contralesional orbit. The pseudo stimulation reproduces during the first and the last 30 seconds of the stimulation, tingling feelings due to current flow experienced during tDCS. In this way there is no possibility for the patient to recognize the difference between the real and the placebo stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Having had a first ischemic stroke within 6 months, or have already had a stroke in the same lesion zone.
* No recurrence.
* Responsible of a right or left hemiplegia.
* Able to walk alone with or without technical assistance.
* Over a distance of at least 10 meters.
* Performance on the six-minute walk test less than 400 meters.
* Without neurological history other than stroke.

Exclusion Criteria:

* Patients who did not have brain MRI after their stroke
* Patients with complete lesion of the primary motor cortex (as identified on MRI).
* Patients with an addiction to alcohol or drugs.
* Patients with psychiatric disease, cognitive impairment disease, uncontrolled epilepsy, neoplastic disease, severe renal or pulmonary failure.
* Patients with cerebellar syndrome associated.
* Patients with clinical involvement of the brainstem (cranial nerve deficit).
* Patients who refused to sign the written consent.
* Patients who have an ongoing pregnancy.
* Patients under justice protection.
* Patients with contraindication to practice aerobic training after stress test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
tDCS tolerance | 2 months
  tolerance questionnaire

SECONDARY OUTCOMES:
Effect size of TDCS on walking performance | 2 months
  Effect size on walking performance (Six-minute walk test (6MWT))

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No